CLINICAL TRIAL: NCT05017688
Title: PrOspective inteRventional Study Exploring the mIcrobiota recolONization in Steroid-Refractory Graft-versus-Host Disease Patients Receiving MaaT013
Brief Title: Prospective Interventional Study Exploring the Microbiota Recolonization in SR-GvHD Patients Receiving MaaT013
Acronym: ORION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MaaT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MPOH07
Record Dates: First submitted 2021-07-09; First posted 2021-08-24 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Intestinal GVHD; Steroid Refractory GVHD
Keywords: gut microbiota; fecal microbiotherapy; intestinal GvHD
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Prospective interventional with low risks and constraints study (RIPH2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient population (Other): The population of the study will be adult patients with GI-aGVHD grade III to IV undergoing MaaT013 treatment through named-patient use program ATUn (Early Access Program).
  Blood and stool samples will be collected at each visit to analyse the gut microbiota and the immune cells.
  Interventions: Procedure: Blood and stool sample collection

INTERVENTIONS:
Procedure: Blood and stool sample collection — Collection of blood samples (55 mL) Collection of fecal samples (10g)

SUMMARY:
The objective of the ORION study is to explore the changes of gut microbiota composition following MaaT013 administration and its impact on the immune system in GVHD patients.

DETAILED DESCRIPTION:
The french regulatory authority ANSM approved in July 2019 the use of MaaT013, a pooled microbiome-based enema formulation, under a formalized named-patient use program in France called "Autorisation Temporaire d'Utilisation - ATU nominative protocolisée - ATUn" or Early Access.

The ATUn is indicated to provide a benefit in the treatment of patients with grade III-IV aGVHD:

* In case of initial resistance to CS alone or in association or in case of failure to other treaments
* In first-line therapy in association with CS in case of steroid-dependance (inability to taper CS dose <0.5 mg/kg/d)
* In case of digestive aGvHD with overlap syndrome The objective of the ORION study is to explore the changes of gut microbiota composition following MaaT013 administration and its impact on the immune system in GVHD patients.

Blood and stool samples will be collected at each visit which explained why the study is thus categorized as research involving the human person with low risks and constraints clinical trial (RIPH2).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old with Grade III-IV aGVHD with gut involvement undergoing treatment with MaaT013 through named-patient use program ATUn / Early Access
* Signature of informed and written consent by the subject or by the subject's legally acceptable representative for patients under guardianship or trusteeship.
* Affiliated or recipient from a social security scheme

Exclusion Criteria:

* Pregnancy and breastfeeding
* Vulnerable patients such as: minors, persons deprived of liberty, persons in Intensive Care Unit unable to provide informed consent prior to the intervention.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of gut microbiota diversity | inclusion (day 0) to month 6
  Diversity of gut microbiota will be evaluated using alpha-diversity metric (Simpson or Shannon or Richness indice) throughout the study
Change of gut microbiota composition | inclusion (day 0) to month 6
  Sample comparisons will be performed using similarity metric such as Bray-Curtis, Jaccard distances, Sorensen, Pearson or Spearman indice.
Change of gut microbiota composition (phylogenetic profiles) | inclusion (day 0) to month 6
  Gut microbiota composition will be evaluated with phylogenetic profiling. Relative abundance of bacterial taxa will be described at each visit throughout the study.

SECONDARY OUTCOMES:
Correlation between gut microbiota and immune parameters | inclusion (day 0) to month 6
  Multiparameter analyses will be performed to identify correlations between changes in gut microbiota composition and immune parameters (Citrulline, Zonulin, ST2, 3 indoxyl sulfate, Reg3a, Total antioxidant status, TGFb1.2.3., IL-1b, IL-2, sIL-2ra, IL-6, IL-8, IL10, IL17-A, IL-18, IFNg, TNFa, sCD14, MCP1, CCL25, CCL28, sCD30, CXCL10)
Gut microbiota baseline characterization based on clinical response | day 0
  Stratification of patients will be based on response to MaaT013 treatment at day 28. Then gut microbiota composition will be described in responder versus non responder patients.
Change in immune parameters following MaaT013 administration | inclusion (day 0) to month 6
  Cytokines and immune parameters of interest (Citrulline, Zonulin, ST2, 3 indoxyl sulfate, Reg3a, Total antioxidant status,TGFb1.2.3., IL-1b, IL-2, sIL-2ra, IL-6, IL-8, IL10, IL17-A, IL-18, IFNg, TNFa, sCD14, MCP1, CCL25, CCL28, sCD30, CXCL10) will be measured in plasma/serum by Luminex and ELISA at each visit and compared to baseline.
  Results will be expressed as ratios on D0 value and heatmap.
  Peripheral blood mononuclear cells will be purified then analyzed by flow cytometry using specific antibodies (CD4, CD8α, CD8β,TCRαβ, CD49a, CCR6, CXCR6, CD25, CD127, CCR7, CD69, CD45RA, CD27, CD57, GITR, CD39, C. Transcriptomic analysis by single cell CITE-seq will be performed on some lymphocytes subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Guenounou, MD, Principal Investigator — IUCT ONCOPOLE
Locations (9):
- France (9):
  - Chu Amiens Picardie Site Sud, Amiens
  - Chu de Caen, Caen
  - Chu Grenoble, Grenoble
  - Chu de Nice - L'Archet 1, Nice
  - Aphp - Hopital Saint Antoine, Paris
  - Chu Lyon Sud, Pierre-Bénite
  - Chu La Miletrie, Poitiers
  - Chu de Rennes - Hopital Pontchaillou, Rennes
  - Institut Universitaire Du Cancer de Toulouse - Oncopole, Toulouse